CLINICAL TRIAL: NCT04786951
Title: AN-VR-ABM: Attentional Bias Modification and Body Exposure Using Virtual Reality and Eye-Tracking to Enhance Treatment for Adolescents With Anorexia Nervosa
Brief Title: Virtual Reality-Based Attention Bias Modification Training for Adolescents With Anorexia Nervosa
Acronym: AN-VR-ABMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, Jose Gutierrez Maldonado, Prof. Dr., University of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2019-108657RB-I00
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: Attentional bias; Virtual Reality; Body exposure procedure; Attentional bias modification training
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Participants were partially randomly assigned to three study groups. To address recruitment challenges due to the limited availability of new adolescent patients and delays in ABMT software development, historical data from a previous randomized controlled trial conducted by the same research team were incorporated. Only participants who met the current study's inclusion and exclusion criteria were included to ensure comparability, as the previous trial employed the same design, assessments, and treatment-as-usual procedures. The historical dataset comprised 21 participants. Newly recruited participants were randomly assigned to one of three groups using block randomization with a computer-generated sequence to ensure balanced group sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual + VR-based body + Attentional Bias Modification Training. (Experimental): In this group, five sessions of VR-based body exposure will be added to the usual treatment, as in the other experimental group. Additionally, at the beginning of each exposure session, participants will undergo attentional bias modification training. The training involves the visual selection of geometric figures that approximately correspond to specific body parts, with each figure presented in different colors. Participants must detect and identify figures appearing on different parts of the avatar's body. In 50% of the trials, discrimination will be based on shape, and in the remaining 50%, it will be based on color. Throughout the training, figures will appear on weight-related body parts in 45% of the trials, on non-weight-related body parts in another 45% of the trials, and on one of three neutral stimuli located next to the avatar in the remaining 10% of trials.
  Interventions: Behavioral: Attentional Bias Modification Training; Behavioral: VR-based body exposure; Behavioral: Usual Care for Eating Disorders
- Treatment as usual + VR-based body exposure (Experimental): Patients assigned to this group will receive the usual treatment provided by their clinical unit, in addition to five weekly sessions of a VR-based body exposure intervention. During these sessions, participants will undergo body exposure using a virtual avatar representing their actual body measurements. The avatar's BMI will be progressively increased across sessions until a healthy BMI is reached.
  Interventions: Behavioral: VR-based body exposure; Behavioral: Usual Care for Eating Disorders
- Treatment as usual (Active Comparator): Patients assigned to this group will receive the usual treatment from the center where they are recruited for the study and will be required to complete the evaluations according to the same schedule as the experimental group.
  Interventions: Behavioral: Usual Care for Eating Disorders

INTERVENTIONS:
Behavioral: Attentional Bias Modification Training — Combine usual treatment with an additional five VR-based body-exposure therapy sessions and five sessions of Attentional Bias Modification Training.
  Arms: Treatment as usual + VR-based body + Attentional Bias Modification Training.
Behavioral: VR-based body exposure — Combine the usual treatment with an additional five VR-based body-exposure therapy sessions
  Arms: Treatment as usual + VR-based body + Attentional Bias Modification Training.; Treatment as usual + VR-based body exposure
Behavioral: Usual Care for Eating Disorders — Participants were recruited from the day-patient and home-treatment programs of the eating disorders unit.
  The day-patient program followed a cognitive-behavioral therapy model and included nutritional rehabilitation, behavioral strategies for improving eating and weight gain, individual and group psychotherapy, and parental support. Attendance ranged from 6 to 11 hours per day, depending on patient risk. The home-treatment program served as transitional care between hospitalization and outpatient treatment and focused on medical stabilization, weight restoration, family involvement, psychoeducation, emotional regulation, and social skills development. Both cognitive-behavioral therapy and family-based therapy were delivered either in person or remotely. Standard treatment procedures for eating disorders were applied across all groups.

SUMMARY:
Anorexia Nervosa (AN) is considered one of the most severe subtypes of eating disorders (EDs), characterized by significant medical complications, high mortality rates, and high comorbidity with other disorders, such as anxiety disorders. Similarly to what occurs in anxiety disorders, several studies have suggested the presence of dysfunctional body-related attentional bias (AB) in patients with EDs, and specifically in patients with AN. Individuals with AN tend to focus their attention on their body in a dysfunctional manner, engaging in body-checking behaviors and excessively scrutinizing their general appearance and weight-related body parts. This body-related AB has been associated with higher levels of body dissatisfaction, which represents one of the most important risk factors for the development and maintenance of EDs.

Moreover, body-related AB may contribute to reducing the effectiveness of body exposure-based treatments used in patients with AN. For this reason, it is necessary to develop new treatment techniques by incorporating specific components aimed at reducing body-related AB. It has been proposed that attentional bias modification techniques could be integrated into body exposure therapy as an effective approach to reduce body-related AB, body dissatisfaction, and body anxiety.

To date, our research group has been the first to use a combination of virtual reality (VR) and eye-tracking (ET) technologies to assess the presence of body-related AB in non-clinical samples. In order to improve treatments for AN, the present project aims to develop a novel attentional bias modification procedure using ET and VR technologies. In addition, this project seeks to integrate this AB modification procedure into a body exposure-based treatment designed to reduce the fear of weight gain experienced by patients with AN.

Finally, the project aims to evaluate whether combining two distinct components-body exposure-based therapy and attentional bias modification training-results in a more effective intervention. It is expected that the inclusion of a VR-based body exposure procedure in standard AN treatment, enhanced through the illusion of ownership over a virtual body, will lead to improved treatment outcomes. Furthermore, it is anticipated that the addition of attentional bias modification training to the body exposure-based procedure will further enhance treatment effectiveness.

DETAILED DESCRIPTION:
Attentional bias (AB) refers to the tendency to allocate greater attention to certain types of stimuli or information (e.g., disorder-relevant information) over other types of information. Adolescent patients with Anorexia Nervosa (AN) have been shown to focus more on self-perceived unattractive body parts than on other body parts. Dysfunctional body-related AB is thought to maintain body image disturbances commonly reported by adolescents with AN by selectively processing body-related information that is consistent with dysfunctional cognitive schemas (e.g., "I am getting a fatter belly"), while schema-inconsistent information (e.g., "I am getting thinner") receives less attention and is often visually neglected.

Dysfunctional body-related AB may also contribute to the reduced effectiveness of body exposure-based treatments for adolescents with AN. Therefore, there is a need to develop novel treatment approaches by incorporating specific components aimed at reducing body-related AB in this population. In a previous project conducted by our group, preliminary evidence supported the effectiveness of body-related AB modification in adolescent patients with AN following a virtual reality (VR)-based mirror exposure intervention. A key factor underlying these results may lie in the structure of the procedure, in which patients were required to sequentially focus on different parts of a virtual body (from head to feet) and verbally express their thoughts and emotions related to each body area.

Building on these findings, the present project aims to further advance this line of research by integrating attentional bias modification techniques into body exposure therapy as an effective approach to reducing body-related AB, body dissatisfaction, and body anxiety in adolescents with AN. To date, our research group has been among the first to combine virtual reality (VR) and eye-tracking (ET) technologies to assess body-related AB in both clinical and non-clinical samples. Specifically, this project seeks to determine whether the addition of attentional bias modification training to body exposure-based therapy results in a more effective intervention for adolescents diagnosed with AN.

It is hypothesized that incorporating AB modification training into the body exposure-based procedure (experimental group) will lead to greater treatment efficacy compared with treatment as usual (control group). Specifically, adolescents in the experimental group are expected to show a significant increase in body mass index (BMI) and a significant reduction in core AN symptomatology (e.g., fear of weight gain, body image disturbances), as well as a reduction in body-related AB, from pre- to post-treatment, compared with the control group. These improvements are also expected to be maintained at the six-month follow-up.

The project will be conducted at the Eating Disorders Units of Hospital Sant Joan de Déu (Barcelona, Spain), which specializes in the treatment of adolescents with eating disorders.

Adolescent patients with AN will be exposed to an immersive virtual environment using a VR head-mounted display (HTC Pro Eye) equipped with integrated eye-tracking. In addition to the two controllers typically provided with the HTC Pro Eye system, three additional body trackers will be used to enable full-body motion tracking. The virtual environment will consist of a room featuring a large mirror positioned on the front wall, approximately 1.5 m in front of the participant, and large enough to reflect the entire body. A young female avatar wearing a basic white T-shirt, blue jeans, and black trainers will be created for the intervention.

Regarding the treatment protocol, all sessions will last approximately one hour and will be conducted once per week. Each session will begin with the induction of the full-body illusion (FBI) and the assessment of visual analogue scales (VASs). Body exposure will initially involve a virtual body with the same BMI as the adolescent patient. The attentional bias modification training will be based on an adaptation of the AB induction procedure proposed by Smeets, Jansen, and Roefs (2011). The training will involve the visual selection of geometric figures (e.g., squares, rectangles, circles) that approximately correspond to specific body parts, with each figure presented in different colors. Participants will be required to detect and identify figures appearing on different parts of the avatar's body. In 50% of the trials, discrimination will be based on shape, while in the remaining 50% it will be based on color. Throughout the training, figures will appear on weight-related body parts in 45% of the trials and on non-weight-related body parts in another 45% of the trials. In the remaining 10% of trials, figures will appear on one of three neutral stimuli positioned next to the avatar.

Raw eye-tracking data will be processed using Ogama (Open Gaze and Mouse Analyzer) software to obtain quantitative measures of visual attention. Weight-related and non-weight-related areas of interest (AOIs) will be defined a priori. Weight-related AOIs will be determined based on the weight-related body items of the PASTAS questionnaire and mapped onto a frontal-view image of a female avatar. These weight-related AOIs will include the legs, thighs, buttocks, hips, abdomen, and waist. All remaining body parts (head, neck, chest, shoulders, arms, and feet) will be classified as non-weight-related AOIs. Selective visual attention will be assessed using total fixation duration and the number of fixations within each AOI.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged 12-17 years.
* Primary diagnosis of anorexia nervosa according to DSM-5 criteria.
* Body weight below the expected range for height, age, and sex.
* Ability to understand and communicate in Spanish.

Exclusion Criteria:

* Presence of severe mental disorders other than anorexia nervosa.
* Significant cognitive impairment that would interfere with participation.
* Visual or auditory deficits that could interfere with VR-based body exposure therapy.
* Epilepsy.
* Pregnancy.
* Cardiac arrhythmia.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Drive for Thinness (EDI-DT) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in drive for thinness scores as measured by the Eating Disorder Inventory-3 - drive for thinness (EDI-DT) scale. Scores range from 0 to 28, with higher scores indicating greater drive for thinness.
Change in Body Dissatisfaction (EDI-BD) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in body dissatisfaction scores as measured by the Eating Disorder Inventory-3 - body dissatisfaction (EDI-BD) scale. Scores range from 0 to 40, with higher scores indicating greater body dissatisfaction.
Change in Body Dissatisfaction (BIAS - BD) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Body dissatisfaction scores were assessed using the Figural Drawing Scale for Body Image Assessment (BIAS-BD). Scores range from -80 to 80, with higher absolute values indicating greater body dissatisfaction.
Change in Body Distortion (BIAS - BD) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Body distortion scores were assessed using the Figural Drawing Scale for Body Image Assessment (BIAS-BD). Scores range from -80 to 80, with higher absolute values indicating greater body distortion.
Change in complete fixation time towards weight-related body parts | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in attentional bias towards weight-related body parts, measured as the total fixation time of gaze (evaluated in milliseconds). Higher values indicate greater attentional bias.
Change in the number of fixations towards weight-related body parts | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in attentional bias towards weight-related body parts, measured as the number of fixations of gaze. Higher values indicate greater attentional bias.
Change in Body Mass Index values | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in Body Mass Index was calculated as weight (kg) divided by height (m) squared. Higher values indicate greater BMI.
Change in Fear of Gaining Weight | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in fear of gaining weight, measured using a visual analogue scale (0-100). Higher scores indicate greater fear of gaining weight.
Change in Anxiety | Assessed at baseline (before the body exposure session); every 2 minutes during the exposure session; at the end of the exposure session; at the end of treatment (6 weeks); and at 6-month follow-up.
  Change in anxiety, measured using a visual analogue scale (0-100). Higher scores indicate greater anxiety.
Change in Body-related Anxiety (PASTAS) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in body-related anxiety as measured by the Physical Appearance State Anxiety Scale (PASTAS). Total scores range from 0 to 32, with higher scores indicating greater body-related anxiety.
Change in Body Appreciation (BAS) | Assessed at baseline, at the end of treatment (6 weeks), and at 6-month follow-up.
  Change in body appreciation as measured by the Body Appreciation Scale (BAS), with scores ranging from 13 to 65; higher scores indicate greater body appreciation.

CONTACTS AND LOCATIONS:
Overall Officials: José Gutiérrez-Maldonado, Principal Investigator — jgutierrezm@ub.edu
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The data presented in this study will be available on request from the corresponding author. The data are not publicly available due to patients' privacy restrictions.

REFERENCES:
- [Background] Reed, D. L., Thompson, J. K., Brannick, M. T., & Sacco, W. P. (1991). Development and validation of the Physical Appearance State and Trait Anxiety Scale (PASTAS). Journal of Anxiety Disorders, 5(4), 323-332. https://doi.org/10.1016/0887-6185(91)90032-O
- [Background] Smeets E, Jansen A, Roefs A. Bias for the (un)attractive self: on the role of attention in causing body (dis)satisfaction. Health Psychol. 2011 May;30(3):360-7. doi: 10.1037/a0022095. PMID 21553980
- [Background] Rodgers RF, DuBois RH. Cognitive biases to appearance-related stimuli in body dissatisfaction: A systematic review. Clin Psychol Rev. 2016 Jun;46:1-11. doi: 10.1016/j.cpr.2016.04.006. Epub 2016 Apr 12. PMID 27116714
- [Background] Bauer A, Schneider S, Waldorf M, Braks K, Huber TJ, Adolph D, Vocks S. Selective Visual Attention Towards Oneself and Associated State Body Satisfaction: an Eye-Tracking Study in Adolescents with Different Types of Eating Disorders. J Abnorm Child Psychol. 2017 Nov;45(8):1647-1661. doi: 10.1007/s10802-017-0263-z. PMID 28133705
- [Background] Tuschen-Caffier B, Bender C, Caffier D, Klenner K, Braks K, Svaldi J. Selective Visual Attention during Mirror Exposure in Anorexia and Bulimia Nervosa. PLoS One. 2015 Dec 29;10(12):e0145886. doi: 10.1371/journal.pone.0145886. eCollection 2015. PMID 26714279
- [Background] Williamson DA, White MA, York-Crowe E, Stewart TM. Cognitive-behavioral theories of eating disorders. Behav Modif. 2004 Nov;28(6):711-38. doi: 10.1177/0145445503259853. PMID 15383683
- [Background] Jansen A, Nederkoorn C, Mulkens S. Selective visual attention for ugly and beautiful body parts in eating disorders. Behav Res Ther. 2005 Feb;43(2):183-96. doi: 10.1016/j.brat.2004.01.003. PMID 15629749